CLINICAL TRIAL: NCT01560624
Title: A Phase III, International, Multi-Center, Randomized, Double-Blind, Placebo-Controlled, Clinical Worsening Study of UT-15C in Subjects With Pulmonary Arterial Hypertension Receiving Background Oral Monotherapy
Brief Title: Phase III Clinical Worsening Study of UT-15C in Subjects With PAH Receiving Background Oral Monotherapy
Acronym: FREEDOM-EV
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: United Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TDE-PH-310
Record Dates: First submitted 2012-03-09; First posted 2012-03-22 (Estimated); Results first posted 2020-02-13 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Pulmonary arterial hypertension (PAH); Pulmonary hypertension (PH); Clinical Worsening; Freedom; Freedom-EV; Treprostinil; UT-15C; 6 Minute walk test
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Hypertension, Pulmonary | interventions — treprostinil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- UT-15C (Experimental): Treprostinil diolamine extended-release tablets (oral) 0.125 to 12 mg TID
  Interventions: Drug: Treprostinil Diolamine
- Placebo (Placebo Comparator): Matching placebo tablets (oral)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Treprostinil Diolamine — Active
  Other Names: UT--15C
  Arms: UT-15C
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is an international, multicenter, randomized, double-blind, placebo-controlled, event driven study in subjects with pulmonary arterial hypertension.

DETAILED DESCRIPTION:
Study TDE-PH-310 is an international, multicenter, randomized (1:1 oral treprostinil (UT-15C): placebo), double-blind, placebo-controlled study in subjects with pulmonary arterial hypertension (PAH) who are receiving background oral monotherapy for PAH for at least 30 days at randomization. Subjects are randomly allocated to receive oral treprostinil extended-release tablets or placebo by a stratified randomization by type of background therapy (Strata 1: phosphodiesterase type 5 inhibitor [PDE5-I] or soluble guanylate cyclase [sGC] stimulator; Strata 2: endothelin receptor antagonist [ERA]. Subjects are also stratified by baseline 6-minute walk distance (6MWD) less than or equal to 350 m or greater than 350 m. Subjects receive their first dose of study drug (0.125 mg) or matching placebo on the day of randomization. Oral dosing of study drug is continued at 0.125 mg 3 times daily (TID; every 6 to 8 hours) with food. The dose (or matching placebo) is titrated throughout the study up to a maximum dose of 12 mg TID to reach and maintain a tolerated dosing regimen that provided optimal clinical benefit. Once randomized, subjects return for study visits every 4 weeks for the first 12 weeks, then every 12 weeks for the duration of the study. Subjects continue in the study until experiencing clinical worsening, the number of adjudicated events necessary for study closure occurr, or prematurely discontinue participation in the study for any reason other than protocol-specified clinical worsening. At each scheduled visit, subjects undergo efficacy assessments for clinical worsening, exercise capacity (6MWD and Borg dyspnea score), WHO functional class (FC), and plasma N-Terminal pro-brain natriuretic peptide (NT-proBNP). Subjects could participate in an optional hemodynamic sub-study (assessed by RHC). Safety assessments consist of adverse events (AEs), physical examinations, vital signs, 12-lead electrocardiograms (ECGs), and clinical laboratory parameters. Patients who complete all required assessments are eligible to enter a long-term, open-label, extension study (TDE-PH-311).

ELIGIBILITY:
Subject Inclusion Criteria:

1. Voluntarily gave informed consent to participate in the study.
2. Are 18 to 75 years of age (inclusive) at Screening.
3. Women of childbearing potential must practice abstinence from intercourse when in line with their preferred and usual lifestyle, or use 2 different forms of highly effective contraception for the duration of the study, and for at least 30 days after discontinuing study medication. A negative urine pregnancy test is required at Screening and Baseline prior to initiating study medication.
4. Male subjects must consent to use a condom during intercourse for the duration of the study, and for at least 48 hours after discontinuing study medication.
5. Have a diagnosis of symptomatic idiopathic or heritable PAH, PAH associated with connective tissue disease (CTD), PAH associated with HIV infection, PAH associated with repaired congenital systemic-to-pulmonary shunt, or PAH associated with appetite suppressant or toxin use.
6. If known to be positive for HIV infection, have a CD4 lymphocyte count of at least 200 cells/mm^3 assessed at Screening and are receiving current standard of care anti retroviral or other effective medication for the treatment of HIV infection.
7. Have a baseline 6MWD greater than or equal to 150 m in the absence of a concurrent injury, illness, or other confounding factor including, but not limited to, use of an aid for ambulation or connection to a nonportable machine, that would have prevented the accurate assessment of the subject's exercise capacity.
8. Are optimally treated with conventional pulmonary hypertension therapy with no additions, discontinuations, or dose changes for a minimum of 10 days prior to randomization. The exceptions are the discontinuation or dose changes of anticoagulants and/or dose change of diuretics.
9. Are receiving a PAH-approved oral monotherapy at a minimum dose that complies with the approved prescribing information for the product for at least 30 days prior to randomization and are receiving a stable dose for at least 10 days prior to randomization.
10. Have had previously undergone a cardiac catheterization within 3 years prior to the start of Screening or during the Screening Period, and the most recent assessment documented a pulmonary artery pressure mean of at least 25 mmHg, a pulmonary capillary wedge pressure (PCWP) (or in the event a PCWP could not be reliably obtained, a left ventricular end diastolic pressure [LVEDP]) less than or equal to 15 mmHg, and absence of unrepaired congenital heart disease (other than patent foramen ovale). If a reliable PCWP or LVEDP are unable to be obtained during cardiac catheterization, subjects with clinically normal left heart function and absence of clinically relevant mitral valve disease on echocardiography are eligible for enrollment.
11. Undergo echocardiography with evidence of clinically normal systolic and diastolic left ventricular function and absence of any clinically significant left sided heart disease (eg, mitral valve disease). Subjects with clinically insignificant left ventricular diastolic dysfunction due to the effects of right ventricular overload (ie, right ventricular hypertrophy and/or dilatation) are eligible.
12. Have a previous ventilation perfusion lung scan, high-resolution computerized tomography scan of the chest, and/or pulmonary angiography that are consistent with the diagnosis of PAH.
13. Have pulmonary function tests conducted within 6 months before Screening or during the Screening Period to confirm the following:

    1. Total lung capacity is at least 60%
    2. Forced expiratory volume at 1 second is at least 50%
14. In the opinion of the Principal Investigator, is able to communicate effectively with study personnel and is considered reliable, willing, and likely to cooperate with protocol requirements, including attending all study visits.

Subject Exclusion Criteria:

1. Is pregnant or lactating.
2. Have previously received oral treprostinil.
3. Have received a PGI2 (except if used during acute vasoreactivity testing) within 30 days prior to randomization or have previous intolerance or significant lack of efficacy to any PGI2 or PGI2 analogue that resulted in discontinuation or inability to titrate that therapy effectively.
4. Have any background conventional therapies for PAH added, removed, or dose-adjusted within 10 days prior to randomization. The exceptions are removal or dose adjustments of anticoagulants and/or dose adjustments of diuretics.
5. Receive their first dose of a PAH-approved oral monotherapy less than 30 days prior to randomization, or have their PAH-approved oral monotherapy dose changed within 10 days prior to randomization, or the subject discontinues any PAH approved therapy within 30 days prior to Screening, or the subject has previously received 2 PAH approved oral therapies at the same time (specifically, a PDE5-I, an ERA, or a sGC stimulator) concomitantly for more than 90 days cumulatively.
6. Have any disease associated with PAH other than CTD, HIV infection, repaired (for at least 1 year) congenital systemic-to-pulmonary shunt, PAH associated with appetite suppressant/toxin use, or have an atrial septostomy.
7. Have a current diagnosis of uncontrolled sleep apnea as defined by their physician.
8. Have a history of ischemic heart disease, including a previous myocardial infarction or symptomatic coronary artery disease within 6 months prior to Screening or a history of left-sided myocardial disease as evidenced by a mean PCWP (or a LVEDP) greater than 15 mmHg or left ventricular ejection fraction less than 40% as assessed by either multigated angiogram, angiography, or echocardiography.
9. Have uncontrolled systemic hypertension as evidenced by systolic blood pressure (BP) greater than 160 mmHg or diastolic BP greater than 100 mmHg.
10. Have alanine aminotransferase or aspartate aminotransferase levels at least 3 times greater than the upper limit of normal, clinically significant liver disease/dysfunction, or known Child-Pugh Class C hepatic disease at Screening.
11. Have any other disease or condition that would interfere with the interpretation of study assessments.
12. Have a musculoskeletal disorder, is using a device to assist walking, or any disease that is likely to limit ambulation, or is connected to a machine that is nonportable.
13. Have an unstable psychiatric condition or is mentally incapable of understanding the objectives, nature, or consequences of the study, or has any condition which in the Investigator's opinion would constitute an unacceptable risk to the subject's safety.
14. Is receiving an investigational drug, have an investigational device in place, or have participated in an investigational drug or device study within 30 days prior to Screening.
15. Have chronic renal insufficiency as defined by either a Screening creatinine value greater than 2.5 mg/dL or the requirement for dialysis.
16. Does not have 3 or more of the following left ventricular disease/dysfunction risk factors:

    1. Body mass index at least 30 kg/m^2
    2. History of essential hypertension
    3. Diabetes mellitus (any type)
    4. Historical evidence of significant coronary artery disease established by any 1 of the following: history of myocardial infarction, percutaneous coronary intervention, or angiographic evidence of coronary artery disease; positive stress test with imaging; previous coronary artery bypass graft; or stable angina.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 690 (Actual)
Dates: Start 2012-06-26 (Actual); Primary Completion 2018-06-24 (Actual); Study Completion 2018-06-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James White, MD, PhD, Principal Investigator — Mary M. Parkes Center
Locations (155):
- United States (40):
  - Arizona Pulmonary Specialists, Ltd., Phoenix, Arizona
  - University of Arizona, Tucson, Arizona
  - University of California, San Francisco-Fresno, Fresno, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California-Davis Medical Group, Advanced Lung Disease/Transplant Program, Sacramento, California
  - David Geffen School of Medicine, Torrance, California
  - University of Colorado Hospital, Aurora, Colorado
  - University of Florida, Gainesville, Florida
  - University of Florida College of Medicine Jacksonville- Division of Pulmonary & Critical Medicine, Jacksonville, Florida
  - University of Florida College of Medicine Jacksonville, Jacksonville, Florida
  - University of Florida College of Medicine, Jacksonville, Jacksonville, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Augusta University, Augusta, Georgia
  - Piedmont - Georgia Lung Associates, Austell, Georgia
  - HeartCare Midwest, Peoria, Illinois
  - Indiana University Hospital, Carmel, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Kentuckiana Pulmonary Associates, Louisville, Kentucky
  - University of Maryland, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Beaumont Health, Troy, Michigan
  - Nebraska Medical Center, Omaha, Nebraska
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - University of Rochester, Rochester, New York
  - Asheville Cardiology Associates, Asheville, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - University Hospital, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Legacy Research Institute, Portland, Oregon
  - Perelman Center for Advanced Medicine; University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center - Presbyterian Cardiovascular Institute, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - Sentara Cardiovascular Research Institute, Norfolk, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
- Argentina (5):
  - Sanatorio San José, CABA, Buenos Aires
  - Hospital Italiano de Buenos Aires, Buenos Aires, Distrito Federal
  - Hospital Italiano Garibaldi, Rosario, Santa Fe Province
  - Sanatorio de la Trinidad Mitre, Buenos Aires
  - Hospital Dr. José María Cullen, Santa Fe
- Australia (8):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Nepean Hospital, Kingswood, New South Wales
  - Saint Vincents Hospital, Sydney, New South Wales
  - Macquarie University, Sydney, New South Wales
  - Prince Charles Hospital, Chermside, Queensland
  - Royal Hobart Hospital, Hobart, Tasmania
  - The Alfred Hospital, Melbourne, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
- Austria (2):
  - Krankenhaus Elisabethinen Linz, Linz, Upper Austria
  - Medizinische Universität Wien, Vienna
- Brazil (8):
  - Hospital das Clinicas da Universidade Federal de Goias, Goiânia, Goiás
  - Hospital das Clínicas da Universidade Federal de Minas Gerais, Belo Horizonte, Minas Gerais
  - Hospital Madre Teresa, Belo Horizonte, Minas Gerais
  - Complexo Hospitalar Santa Casa de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital das Clínicas da Faculdade de Medicina de Botucatu- UNESP, Botucatu, São Paulo
  - Hospital da Clínicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo, São Paulo
  - Escola Paulista de Medicina, Universidade Federal de São Paulo, São Paulo, São Paulo
  - Hospital Alemão Oswaldo Cruz, São Paulo
- Canada (4):
  - Respiratory Research Foundation, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Vancouver Coastal Health, Vancouver, British Columbia
  - Lawson Health Research Institute, London, Ontario
- Chile (2):
  - Centro de Investigaciones TASOL, Santiago, Santiago Metropolitan
  - Clínica Tabancura, Vitacura, Santiago Metropolitan
- China (16):
  - Beijing Chao-Yang Hospital, Beijing, Beijing Municipality
  - Guangdong General Hospital, Guangzhou, Guangdong
  - Wuhan Asia Heart Hospital, Wuhan, Hubei
  - Xiangya Hospital, Changsha, Hunan
  - The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - The Second Affiliated Hospital of Nanchang Medical University, Nanchang, Jiangxi
  - Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality
  - Renji Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - West China Hospital, Chengdu, Sichuan
  - Peking Union Medical College Hospital, Beijing
  - Beijing Shijitan Hospital, Beijing
  - Chinese PLA General Hospital, Beijing
  - The Affiliated Hospital of Qingdao University, Qingdao
  - Renji Hospital of Shanghai Jiaotong University, Shanghai
  - Shanghai Pulmonary Hospital of Tongji University, Shanghai
  - Shenyang General Hospital of Shenyang Military Command, Shenyang
- Denmark (2):
  - Aarhus Universitetshospital, Skejby, Aarhus
  - Rigshospitalet-Copenhagen University Hospital, Copenhagen
- France (6):
  - Hopital Haut-Leveque, CHU Bordeaux, Pessac, Aquitaine
  - Hopital Jean Minjoz Centre Hospitalier Universitaire Besancon, Besançon, Franche-comte
  - Centre Hospitalier Régional Universitaire de Lille - Hôpital Claude Huriez, Lille, Hauts-de-France
  - CHU de Montpellier, Montpellier, Languedoc-roussillon
  - Hopital Brabois, Vandœuvre-lès-Nancy, Limousin, Lorraine
  - Centre Hospitalier Universitaire Hopital Nord, Marseille, Provence-Alpes-Côte d'Azur Region
- Germany (14):
  - Thoraxklinik am Universitätsklinikum Heidelberg, Heidelberg, Baden-Wurttemberg
  - Ludwig-Maximilians-Universitat Munchen, München, Bavaria
  - Universitätsklinikum Regensburg, Regensburg, Bavaria
  - Missionsarztliche Klinik Wurzburg gGmbH, Würzburg, Bavaria
  - Universitätsmedizin Greifswald, Greifswald, Mecklenburg-Vorpommern
  - Bergmannsheil Berufsgenossenschaftliche Universitätsklinik GmbH, Bochum, North Rhine-Westphalia
  - Universitätsklinikum Köln, Cologne, North Rhine-Westphalia
  - Herzzentrum Duisburg, Duisburg, North Rhine-Westphalia
  - Universitätsmedizin der Johannes Gutenberg Universität, Mainz, Rhineland-Palatinate
  - Universitätsklinikum des Saarlandes, Homburg, Saarland
  - Technische Universität Dresden, Dresden, Saxony
  - Universitätsklinikum Leipzig, Leipzig, Saxony
  - Universitätskrankenhaus Hamburg-Eppendorf, Hamburg
  - Technische Universität Dresden, Sachsen
- Greece (2):
  - University General Hospital of Attikon, Athens, Attica
  - General Hospital of Thessaloniki, "G.Papanikolaou", Thessaloniki, Macedoni
- India (12):
  - CARE Hospital, Hyderabad, Andhra Pradesh
  - Mediciti Hospital, Hyderabad, Andhra Pradesh
  - Care Institute Medical Sciences, Ahmedabad, Gujarat
  - Apollo Hospitals International, Ltd., Gandhinagar, Gujarat
  - Medanta - The Medicity, Gurgaon, Haryana
  - Narayana Institute of Cardiac Sciences, Bangalore, Karnataka
  - KEM Hospital, Mumbai, Maharashtra
  - Ruby Hall Clinic, Pune, Maharashtra
  - Sir Ganga Ram Hospital, New Delhi, National Capital Territory of Delhi
  - Indraprastha Apollo Hospital, New Delhi, National Capital Territory of Delhi
  - Apollo Hospital, Chennai, Tamil Nadu
  - G. Kuppuswamy Naidu Memorial Hospital, Coimbatore, Tamil Nadu
- Israel (5):
  - Rabin Medical Center, Petach Tikvah, Petah Tiqwa
  - The Chaim Sheba Medical Center at Tel Hashomer, Tel Litwinsky, Tel Aviv
  - Rambam Health Corp., Haifa
  - Carmel Medical Center, Haifa
  - Hadassah Medical Center, Jerusalem
- Italy (4):
  - Azienda Ospedaliera Universitaria, Napoli
  - Istituto Mediterraneo Trapianti e Terapia Alta Specializzazione (ISMETT), Palermo
  - Fondazione IRCCS Policlinico S. Matteo, Pavia
  - Azienda Policlinico Umberto I di Roma, Roma
- Mexico (2):
  - Instituto Nacional de Cardiologia Ignacio Chavez, Tlalpan, Mexico City
  - Unidad de Investigacion Clinica en Medicina S.C., Monterrey, Nuevo León
- Netherlands (2):
  - Universitair Medisch Centrum Sint Radboud, Nijmegen, Gelderland
  - Vrije Universiteit Medisch Centrum, Amsterdam, North Holland
- Poland (4):
  - Uniwersytecki Szpital Kliniczny w Bialymstoku, Bialystok
  - Szpital Kliniczny Przemienienia Panskiego Uniwersytetu Medycznego im K. Marcinkowskiego w Poznaniu, Krakow
  - Krakowski Szpital Specjalistyczny im. Jana Pawla II, Małogoskie
  - Europejskie Centrum Zdrowia Otwock, Szpital im. Fryderyka Chopina, Otwock
- Singapore (2):
  - National University Hospital, Singapore
  - National Heart Centre Singapore, Singapore
- South Korea (5):
  - Gachon University Gil Medical Center, Incheon
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul
  - Asan Medical Center, Seoul
- Sweden (2):
  - Sahlgrenska University Hospital, Gothenburg, Västra Götaland County
  - Karolinska University Hospital Solna, Stockholm
- Taiwan (4):
  - National Cheng Kung University Hospital, Tainan, Tainan CITY
  - Veterans General Hospital-Kaohsiung, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
- United Kingdom (4):
  - Papworth Hospital, Papworth Everard, Cambridgshire
  - Royal Free Hospital, London, England
  - Freeman Hospital, Newcastle upon Tyne, England
  - Royal Hallamshire Hospital, Sheffield, England

REFERENCES:
- [Derived] White RJ, Jerjes-Sanchez C, Bohns Meyer GM, Pulido T, Sepulveda P, Wang KY, Grunig E, Hiremath S, Yu Z, Gangcheng Z, Yip WLJ, Zhang S, Khan A, Deng CQ, Grover R, Tapson VF; FREEDOM-EV Investigators. Combination Therapy with Oral Treprostinil for Pulmonary Arterial Hypertension. A Double-Blind Placebo-controlled Clinical Trial. Am J Respir Crit Care Med. 2020 Mar 15;201(6):707-717. doi: 10.1164/rccm.201908-1640OC. PMID 31765604

RESULTS

PARTICIPANT FLOW:
Groups:
- UT-15C: Treprostinil diolamine extended-release tablets (oral) 0.125 to 12 mg three times daily (TID)
  Treprostinil Diolamine: Active
Period: Overall Study
Arm/Group | UT-15C | Placebo
Started | 346 | 344
Clinical Worsening Event (Including death) | 91 | 133
Early Discontinuation From Treatment (Due to progressive disease, AE, withdrawal by subject, protocol violation, lost to follow-up) | 107 | 56
Completed (Completed the study without clinical worsening or early discontinuation) | 148 | 155
Not Completed | 198 | 189

BASELINE CHARACTERISTICS:
Population: The Intent-to-Treat (ITT) Population was defined as all subjects randomized into the study who received at least 1 dose of study drug. The Safety Population was defined as all subjects in the study that received study drug. ITT subjects with major protocol deviations were excluded from the Per-Protocol population.
Groups:
- Total: Total of all reporting groups
Arm/Group | UT-15C | Placebo | Total
Number analyzed (Participants) | 346 | 344 | 690
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 292 | 294 | 586
  >=65 years | 54 | 50 | 104
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.6 (15.7) | 44.8 (15.4) | 45.2 (15.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 275 | 269 | 544
  Male | 71 | 75 | 146
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 150 | 156 | 306
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 13 | 21
  White | 187 | 173 | 360
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  North America | 39 | 54 | 93
  Southeast Asia | 162 | 160 | 322
  Europe | 55 | 44 | 99
  South America | 90 | 86 | 176
Time since Diagnosis [Mean (Standard Deviation); unit: years] | 1.34 (2.50) | 1.37 (2.58) | 1.35 (2.54)
6MWD at Baseline [Mean (Standard Deviation); unit: meters] | 392.9 (92.5) | 398.5 (100.0) | 395.7 (96.3)
Etiology of PAH [Count of Participants; unit: Participants]
  Idiopathic or Heritable PAH | 219 | 216 | 435
  Collagen Vascular Disease | 94 | 84 | 178
  HIV Infection | 2 | 7 | 9
  Congenital Heart Defect | 20 | 27 | 47
  Other | 11 | 10 | 21
WHO Functional Class at Baseline [Count of Participants; unit: Participants] — WHO FC I describes patients who do not experience symptoms with exercise or at rest. WHO FC II describes patients who experience symptoms with ordinary activities but not at rest. WHO FC III describes patients who are limited in normal activities but do not experience symptoms at rest. WHO FC IV describes patients who are symptomatic at rest and experience severe symptoms with any activity.
  Participants
    I | 9 | 13 | 22
    II | 205 | 228 | 433
    III | 131 | 103 | 234
    IV | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Time to First Clinical Worsening Event
Description: Clinical worsening was assessed continuously from randomization until the subject's last study visit. Clinical worsening events were defined as death (all causes), hospitalizations due to worsening pulmonary arterial hypertension (PAH), initiation of an inhaled or infused prostacyclin (PGI2) for the treatment of worsening PAH, disease progression, or unsatisfactory long-term clinical response. All clinical worsening events reported by the study sites were reviewed by the Sponsor Medical Monitors. Once a clinical worsening event occurred, it was entered in the eCRF and a narrative was submitted for review by the Sponsor's Medical Monitor within 48 hours after the event became known to the Investigator or designee. Subsequently, the narratives for subjects with the reported clinical worsening events were sent to an independent adjudication committee. The independent adjudication committee reviewed and adjudicated all clinical worsening events throughout the study.
Time Frame: From randomization to approximately 4 years
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | UT-15C | Placebo
Number analyzed (Participants) | 346 | 344
weeks | 60.58 (42.93) | 49.31 (46.28)
Statistical Analysis 1: Comparison: UT-15C vs Placebo; Test type: Superiority; p = 0.0275, Cox proportion-hazard model; Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.56 to 0.97]
Statistical Analysis 2: Comparison: UT-15C vs Placebo; Test type: Superiority; p = 0.0391, Log Rank

2. Secondary Outcome: Change in 6-Minute Walk Distance
Description: The intent of the 6-Minute Walk Test (6MWT) is to evaluate exercise capacity associated with carrying out activities of daily living. A baseline 6MWT was performed prior to initiation of study drug on the day of randomization. 6MWTs were conducted at Weeks 4, 8, 12, 24, and every 12 weeks thereafter. The change between Baseline and Week 24 is reported.
Time Frame: From Baseline to Week 24
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | UT-15C | Placebo
Number analyzed (Participants) | 346 | 344
meters
  Baseline | 392.9 (92.5) | 398.5 (100.00)
  Week 24 | 395.4 (120.0) | 372.3 (163.0)
Statistical Analysis 1: Comparison: UT-15C vs Placebo; Test type: Superiority; p = 0.0913, ANCOVA; Hodges Lehmann estimate location shift = 7.0, 95% CI 2-sided [0 to 16.0]

3. Secondary Outcome: Change in Plasma N-Terminal Pro-brain Natriuretic Peptide (NT-proBNP) From Baseline to Week 24
Description: Plasma NT-proBNP concentration is a useful biomarker for the severity of PAH as it is associated with changes in right heart morphology and function. NT-proBNP sample collection occurred at Baseline (prior to starting study drug), Week 12, Week 24, the first Continued Visit, and every other Continued Visit thereafter (ie, Continued Visits 3, 5, 7, etc). NT-proBNP was also assessed at the Study Drug Termination Visit. The change between Baseline and Week 24 is reported.
Time Frame: From Baseline to Week 24
Population: Subjects who did not have a valid NT-proBNP measurement at Baseline or Week 24 were excluded from the analysis.
Measure: Least Squares Mean (Standard Error); unit: Ratio to baseline
Arm/Group | UT-15C | Placebo
Number analyzed (Participants) | 346 | 344
Ratio to baseline | 0.7859 (1.05470) | 1.1230 (1.05439)
Statistical Analysis 1: Comparison: UT-15C vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA

4. Secondary Outcome: Change in World Health Organization Functional Class (WHO FC) From Baseline to Week 48
Description: The WHO FC for PAH was assessed at Baseline prior to starting study drug, at all subsequent scheduled study visits, and every time the 6MWT was performed for purposes of assessing clinical worsening status.
Time Frame: Baseline to Week 48
Measure: Count of Participants; unit: Participants
Arm/Group | UT-15C | Placebo
Number analyzed (Participants) | 315 | 311
Participants
  Improved | 46 | 38
  No change | 203 | 170
  Deteriorated | 66 | 103
Statistical Analysis 1: Comparison: UT-15C vs Placebo; Test type: Superiority; p = 0.0028, Fisher Exact

ADVERSE EVENTS:
Time Frame: The study lasted 6 years; however, subjects remained in the study for various durations. The longest subject duration in the study was 5.1 years.
Arm/Group | UT-15C | Placebo
All-Cause Mortality (participants affected / at risk) | 17/346 | 18/344
Serious Adverse Events (participants affected / at risk) | 116/346 | 110/344
Other Adverse Events (participants affected / at risk) | 342/346 | 328/344
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | UT-15C (N=346) | Placebo (N=344)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 26 (27) | 36 (40)
Right ventricular failure (Cardiac disorders) | 17 (18) | 12 (12)
Pneumonia (Infections and infestations) | 10 (11) | 10 (11)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 8 (9)
Cardiac failure (Cardiac disorders) | 5 (5) | 3 (3)
Gastroenteritis (Infections and infestations) | 5 (5) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 5 (5) | 3 (3)
Bronchitis (Infections and infestations) | 4 (4) | 3 (3)
Headache (Nervous system disorders) | 4 (4) | 2 (2)
Lung infection (Infections and infestations) | 4 (4) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Septic shock (Infections and infestations) | 3 (3) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 2 (2)
Appendicitis (Infections and infestations) | 2 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 1 (1)
Chest discomfort (General disorders) | 2 (2) | 0 (0)
Chest pain (General disorders) | 2 (2) | 5 (5)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
Circulatory collapse (Vascular disorders) | 2 (2) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Gastritis erosive (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 2 (2) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 4 (5)
Lower respiratory tract infection (Infections and infestations) | 2 (2) | 2 (2)
Sudden death (General disorders) | 2 (2) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 4 (4)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (2) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0)
Acute lung injury (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (5)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arteriovenous malformation (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Asthenia (General disorders) | 1 (1) | 2 (2)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Brain injury (Nervous system disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 3 (3)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 2 (2)
Cardio-respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 4 (4)
Cardiovascular insufficiency (Cardiac disorders) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 0 (0)
Catheterisation cardiac (Investigations) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Cor pulmonale (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticulum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal ulcer haemorhage (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Emotional distress (Psychiatric disorders) | 1 (1) | 0 (0)
Erosive duodenitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Femoral vein perforation (Vascular disorders) | 1 (1) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Foetal death (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal bacterial (Infections and infestations) | 1 (1) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Glomerulonephritis rapidly progressive (Renal and urinary disorders) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (4)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hepatic cyst (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypovolaemic shock (Vascular disorders) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 2 (2)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Nephrotic syndrome (Renal and urinary disorders) | 1 (1) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Ovarian rupture (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Oxygen saturation decreased (Investigations) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Palatal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 4 (4)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 4 (4)
Shock haemorrhagic (Vascular disorders) | 1 (1) | 0 (0)
Sinus node dysfunction (Cardiac disorders) | 1 (1) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Tracheobronchitis (Infections and infestations) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Uterine cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Uterine tumour excision (Surgical and medical procedures) | 1 (1) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Adjustment disorder with depressed mood (Psychiatric disorders) | 0 (0) | 1 (1)
Altered state of consciousness (Psychiatric disorders) | 0 (0) | 1 (1)
Appendiceal abscess (Infections and infestations) | 0 (0) | 1 (1)
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ascites (Cardiac disorders) | 0 (0) | 1 (1)
Atypical pneumonia (Infections and infestations) | 0 (0) | 1 (2)
Autoimmune hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Chronic gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1)
Chronic sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Dengue fever (Infections and infestations) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Exostosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Gastrointestinal angiodysplasia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hepatic cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (3)
Hepatic mass (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Implant site irritation (General disorders) | 0 (0) | 1 (1)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 (0) | 1 (1)
Incarcerated umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 1 (1)
Inguinal hernia strangulated (Gastrointestinal disorders) | 0 (0) | 1 (1)
Interleukin level increased (Investigations) | 0 (0) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 1 (1)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Oedema peripheral (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Optic neuritis (Nervous system disorders) | 0 (0) | 1 (1)
Organising pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Panniculitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 2 (2)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal transplant (Surgical and medical procedures) | 0 (0) | 1 (1)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Retinal vein occlusion (Eye disorders) | 0 (0) | 1 (1)
Scleroderma renal crisis (Renal and urinary disorders) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal decompression (Surgical and medical procedures) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Vocal cord paresis (Nervous system disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | UT-15C (N=346) | Placebo (N=344)
Anaemia (Blood and lymphatic system disorders) | 17 (17) | 12 (17)
Palpitations (Cardiac disorders) | 47 (48) | 31 (35)
Right ventricular failure (Cardiac disorders) | 22 (23) | 19 (19)
Diarrhoea (Gastrointestinal disorders) | 240 (277) | 98 (106)
Nausea (Gastrointestinal disorders) | 139 (146) | 78 (90)
Vomiting (Gastrointestinal disorders) | 123 (135) | 35 (37)
Abdominal pain upper (Gastrointestinal disorders) | 40 (41) | 17 (20)
Abdominal discomfort (Gastrointestinal disorders) | 29 (30) | 12 (14)
Abdominal pain (Gastrointestinal disorders) | 28 (30) | 13 (13)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 24 (25) | 12 (12)
Abdominal distension (Gastrointestinal disorders) | 27 (28) | 16 (16)
Dyspepsia (Gastrointestinal disorders) | 18 (19) | 20 (20)
Constipation (Gastrointestinal disorders) | 16 (18) | 9 (10)
Gastritis (Gastrointestinal disorders) | 16 (16) | 7 (8)
Oedema peripheral (General disorders) | 46 (50) | 81 (89)
Fatigue (General disorders) | 37 (43) | 46 (48)
Chest discomfort (Gastrointestinal disorders) | 29 (32) | 30 (32)
Chest pain (General disorders) | 26 (34) | 45 (48)
Pyrexia (General disorders) | 25 (26) | 26 (28)
Aesthenia (General disorders) | 23 (23) | 17 (18)
Oedema (General disorders) | 17 (17) | 12 (12)
Upper respiratory tract infection (Infections and infestations) | 73 (105) | 82 (109)
Viral upper respiratory tract infection (Infections and infestations) | 56 (69) | 46 (63)
Bronchitis (Infections and infestations) | 24 (27) | 19 (25)
Pneumonia (Infections and infestations) | 16 (18) | 17 (18)
Urinary tract infection (Infections and infestations) | 16 (20) | 17 (20)
Influenza (Infections and infestations) | 13 (13) | 17 (18)
Decreased appetite (Metabolism and nutrition disorders) | 32 (33) | 16 (16)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 62 (64) | 10 (11)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 61 (78) | 30 (32)
Myalgia (Musculoskeletal and connective tissue disorders) | 49 (53) | 37 (42)
Arthralgia (Musculoskeletal and connective tissue disorders) | 41 (51) | 31 (39)
Back pain (Musculoskeletal and connective tissue disorders) | 31 (32) | 27 (27)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 10 (12) | 22 (23)
Headache (Nervous system disorders) | 259 (283) | 120 (134)
Dizziness (Nervous system disorders) | 81 (86) | 75 (83)
Syncope (Nervous system disorders) | 20 (23) | 20 (24)
Insomnia (Psychiatric disorders) | 22 (22) | 16 (17)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 56 (61) | 77 (88)
Cough (Respiratory, thoracic and mediastinal disorders) | 46 (48) | 63 (72)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 38 (39) | 64 (70)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 21 (25) | 31 (33)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 20 (21) | 17 (19)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 18 (19)
Rash (Skin and subcutaneous tissue disorders) | 19 (19) | 15 (17)
Flushing (Vascular disorders) | 154 (158) | 27 (28)
Hypotension (Vascular disorders) | 24 (24) | 14 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution and/or Principal Investigator agree not to publish or publicly present any interim results of the Study without the prior written consent of Sponsor, not to be unreasonably withheld or delayed. Institution and/or Principal Investigator further agree to provide Sponsor with drafts of any such publication or presentation for review and approval no less than 30 days prior to submission for publication or the date of public presentation.

DOCUMENTS (2):
  • Study Protocol (2017-08-09): https://cdn.clinicaltrials.gov/large-docs/24/NCT01560624/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-08): https://cdn.clinicaltrials.gov/large-docs/24/NCT01560624/SAP_001.pdf